CLINICAL TRIAL: NCT02832258
Title: Urinary Tract Infection Due to Extended-spectrum Beta-lactamase-producing Enterobacteriaceae in Children: an Observational French Study
Brief Title: Urinary Tract Infection Due to Beta-lactamase-producing Enterobacteriaceae in Children
Acronym: PYELOBLSE
Status: Completed | Type: Observational
Sponsor: Fouad Madhi (Other)
Responsible Party: Sponsor-Investigator, Fouad Madhi, Dr, Centre Hospitalier Intercommunal Creteil
Organization: Centre Hospitalier Intercommunal Creteil (Other)
Other Study IDs: PYELOBLSE
Record Dates: First submitted 2016-06-29; First posted 2016-07-14 (Estimated); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Urinary Tract Infections
Keywords: Enterobacteria; Children; Febrile urinary tract infection; Cystitis; Extended-spectrum beta-lactamase-producing Enterobacteriaceae
MeSH Terms: conditions — Urinary Tract Infections; Cystitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children with urinary tract infection due to E-ESBL: In this prospective observational study between March 2013 and March 2017, children (0 to 18 years) with E-ESBL UTI (febrile UTI or cystitis) were enrolled in 24 pediatric departments in France. Clinical and biological characteristics, risk factors of infection of E-ESBL, first and second lines of antibiotic therapies were analyzed. We used the Kaplan-Meier method to estimate the time to apyrexia and length of hospital stay, and Log-rank test to assess equality of survivor functions. We also analyzed the resistance patterns and molecular characterization of ESBL types in the isolates.

SUMMARY:
Urinary tract infection due to Extended-spectrum beta-lactamase producing enterobacteriaceae (E-ESBL UTI) become a frequent problem. A too large variety in the prescription of antibiotics for E-ESBL UTI in children and absolute recommendations regarding the optimal treatment of E-ESBL is nearly impossible at this time.

Our aim was to describe the characteristics and treatments of urinary tract infections caused by Extended spectrum betalactamase-producing Enterobacteriaceae in children.

DETAILED DESCRIPTION:
In this prospective observational study between March 2013 and March 2017, children (0 to 18 years) with ESBL-E UTI were enrolled in 24 pediatric departments in France. Clinical and biological characteristics, risk factors of infection of E-ESBL, first and second lines of antibiotic therapies were analyzed. The investigators used the Kaplan-Meier method to estimate the time to fever defervescence and hospitalization duration, and Log-rank test to assess equality of survivor functions. The investigators also analyzed the resistance patterns and molecular characterization of ESBL types in the isolates.

ELIGIBILITY:
Inclusion Criteria:

* All inpatient or outpatient under 18 years with UTI (cystitis or febrile UTI)
* Clinical signs associated with a positive E-ESBL in urine culture dependent urine collection method as previously described (Stein R, EAU/ESPU guidelines) and an antibiotic treatment targeting this strain.

Exclusion Criteria:

* Refusal to participate in the study
* Children with mixed microbial strains and repeated infections were excluded

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study was created by the GPIP/ACTIV network with 24 pediatric centers (pediatric and emergency department) working with their microbiology departments throughout France. Between March 2014 and March 2017, they enrolled all children treated for UTI by E-ESBL in this prospective observational study. These hospitals were located in 7 regions (Ile de France, Nord-Pas-de-Calais-Picardie, Provence-Alpes-Côte d'Azur, Seine-Maritime, Rhône and Loire-Atlantique). For this hospital-based active surveillance, a clinical investigator in each participating ward completed a standardized data form sent by electronic or postal mail to the investigating center. All data were validated by a scientific committee.
Sampling Method: Non-Probability Sample
Enrollment: 590 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
First and second lines used antibiotic therapies | at inclusion, at 3 days

SECONDARY OUTCOMES:
Resistance patterns of ESBL types in the isolates | at inclusion
  On the fisrt hundred urine samples
Clinical characteristics (fewer, clinical sepsis) of E-ESBL UTI in children | at inclusion
Time to apyrexia (Kaplan-Meier method) | at inclusion
Length of hospital stay (Kaplan-Meier method) | at inclusion
Molecular characterization of ESBL types in the isolates | at inclusion
  On the fisrt hundred urine samples
Clinical history of patient with E-ESBL UTI in children | at inclusion
C reactive protein level of patient with E-ESBL UTI in children | at inclusion
procalcitonin level of patient with E-ESBL UTI in children | at inclusion
Positive blood culture | at inclusion
cytobacteriological examination of the urine results | at inclusion, at 3 days
urine analysis by regent strip method | at inclusion

CONTACTS AND LOCATIONS:
Locations (24):
- France (24):
  - Hopital Ambroise Paré, Boulogne-Billancourt
  - Saint Camille Hospital, Bry-sur-Marne
  - Louis Mourier Hospital, Colombes
  - CHI Créteil, Créteil
  - Centre Hospitalier de Dourdan, Dourdan
  - CHU Le Havre, Le Havre
  - CHU Le Kremlin-Bicêtre, Le Kremlin-Bicêtre
  - Roger Salengro Hospital, Lille
  - Centre Hospitalier Général de Longjumeau, Longjumeau
  - CHU Lyon, Lyon
  - Centre Hospitalier de Meaux, Meaux
  - Centre Hospitalier Marc Jacquet, Melun
  - CHU Nantes, Nantes
  - CHU Lenval, Nice
  - Centre Hospitalier d'Orsay, Orsay
  - Hospital Trousseau, Paris
  - Hôpital Necker, Paris
  - Robert Debré, Paris
  - Centre Hospitalier Roubaix, Roubaix
  - CHU Rouen, Rouen
  - Hôpital Intercommunal de Villeneuve Saint-Georges, Villeneuve-Saint-Georges
  - Jean Verdier Hospital, Bondy, Île-de-France Region
  - Antoine Beclère Hospital, Clamart, Île-de-France Region
  - André Mignot Hospital, Le Chesnay, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng CH, Tsai MH, Huang YC, Su LH, Tsau YK, Lin CJ, Chiu CH, Lin TY. Antibiotic resistance patterns of community-acquired urinary tract infections in children with vesicoureteral reflux receiving prophylactic antibiotic therapy. Pediatrics. 2008 Dec;122(6):1212-7. doi: 10.1542/peds.2007-2926. PMID 19047236
- [Background] Paterson DL, Ko WC, Von Gottberg A, Mohapatra S, Casellas JM, Goossens H, Mulazimoglu L, Trenholme G, Klugman KP, Bonomo RA, Rice LB, Wagener MM, McCormack JG, Yu VL. Antibiotic therapy for Klebsiella pneumoniae bacteremia: implications of production of extended-spectrum beta-lactamases. Clin Infect Dis. 2004 Jul 1;39(1):31-7. doi: 10.1086/420816. Epub 2004 Jun 8. PMID 15206050
- [Background] Boyer-Mariotte S, Duboc P, Bonacorsi S, Lemeland JF, Bingen E, Pinquier D. CTX-M-15-producing Escherichia coli in fatal neonatal meningitis: failure of empirical chemotherapy. J Antimicrob Chemother. 2008 Dec;62(6):1472-4. doi: 10.1093/jac/dkn362. Epub 2008 Sep 4. No abstract available. PMID 18772159
- [Background] Fournier S, Brun-Buisson C, Jarlier V. Twenty years of antimicrobial resistance control programme in a regional multi hospital institution, with focus on emerging bacteria (VRE and CPE). Antimicrob Resist Infect Control. 2012 Feb 13;1(1):9. doi: 10.1186/2047-2994-1-9. PMID 22958336
- [Background] Birgy A, Cohen R, Levy C, Bidet P, Courroux C, Benani M, Thollot F, Bingen E. Community faecal carriage of extended-spectrum beta-lactamase-producing Enterobacteriaceae in French children. BMC Infect Dis. 2012 Nov 21;12:315. doi: 10.1186/1471-2334-12-315. PMID 23171127
- [Background] Madec JY, Lazizzera C, Chatre P, Meunier D, Martin S, Lepage G, Menard MF, Lebreton P, Rambaud T. Prevalence of fecal carriage of acquired expanded-spectrum cephalosporin resistance in Enterobacteriaceae strains from cattle in France. J Clin Microbiol. 2008 Apr;46(4):1566-7. doi: 10.1128/JCM.02299-07. Epub 2008 Feb 13. No abstract available. PMID 18272707
- [Background] Andriatahina T, Randrianirina F, Hariniana ER, Talarmin A, Raobijaona H, Buisson Y, Richard V. High prevalence of fecal carriage of extended-spectrum beta-lactamase-producing Escherichia coli and Klebsiella pneumoniae in a pediatric unit in Madagascar. BMC Infect Dis. 2010 Jul 12;10:204. doi: 10.1186/1471-2334-10-204. PMID 20624313